CLINICAL TRIAL: NCT01556880
Title: A Randomized Controlled Trial of Short Message Service by Cellular Phone for Professional Drivers With Pre-diabetes
Brief Title: RCT of SMS for Drivers With Pre-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Eastern Hospital (Unknown)
Responsible Party: Principal Investigator, WONG King Ho Carlos, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HKCTR-560
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Pre-diabetes; Diabetes
Keywords: Drivers; Chinese; Short Message Service; Cellular Phone
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Message Service (SMS) (Experimental): A computer-based text message database was created. Messages prompted subjects to get rid of smoking and eating out, to persevere with the quit smoking attempt with the emphasis on the peer pressure on the smoking cessation by the smoking ban in restaurants. They encouraged them to overcome the barriers of healthy eating diet and physical activity with a block of text messages.
  Interventions: Behavioral: Short Message Service (SMS)
- Standard usual care (No Intervention)

INTERVENTIONS:
Behavioral: Short Message Service (SMS) — A computer-based text message database was created. Messages prompted subjects to get rid of smoking and eating out, to persevere with the quit smoking attempt with the emphasis on the peer pressure on the smoking cessation by the smoking ban in restaurants. They encouraged them to overcome the barriers of healthy eating diet and physical activity with a block of text messages.
  Arms: Short Message Service (SMS)

SUMMARY:
The purpose of this study is to prevent the professional drivers from pre-diabetes to diabetes.

DETAILED DESCRIPTION:
Mobile phone use is almost a routine part of society worldwide. All mobile phones can deliver and receive short-messaging service text messages, providing a perfect medium for delivering information and support. Since short-messaging service is little exploited in clinical research or practice in Chinese population, this study examined the effectiveness of one-way messaging which is less expensive and is easier to undertake. We aimed to determine the effectiveness of using SMS to provide pre-diabetes and diabetes information by promoting healthy lifestyle modification and reducing the two-hour post-glucose loading plasma glucose, the risk of acquiring Type 2 Diabetes Mellitus among professional drivers with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* identified within the last 3 months with pre-diabetes which is defined as a fasting plasma glucose level of 5.6-6.9 mmol/L or a two-hour level after a 75 grams glucose load of 7.8-11 mmol/L based on the World Health Organization 1998 criteria;
* accessible by mobile phone that could receive Chinese text messages.

Exclusion Criteria:

* a history of diabetes mellitus;
* currently on medicines known to alter glucose tolerance;
* did not have a mobile phone;
* unable to read Chinese characters;
* refused to take part in current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
incidence rate of DM | Follow-up in 12 months
  the incidence rate of DM during first year 12-month period

SECONDARY OUTCOMES:
Body mass index | Baseline, follow-up in 12 months and 24 months
Waist Circumference | Baseline, follow-up in 12 months and 24 months
Fasting Glucose | Baseline, follow-up in 12 months and 24 months
  Fasting plasma glucose and two-hour post-meal loading plasma glucose
Blood pressure | Baseline, follow-up in 12 months and 24 months
  Systolic blood pressure and diastolic blood pressure
Lipid profile | Baseline, follow-up in 12 months and 24 months
  Total cholesterol, triglycerides, high density lipoprotein cholesterol and low density lipoprotein cholesterol
incidence of DM | Follow-up in 24 months
  incidence of DM for first two year 24-month period

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, The University of Hong Kong; Yvonne Y.C. Lo, MBBS, Principal Investigator — Department of Family Medicine and Primary Care, The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Department of Family Medicine and Primary Care, The University of Hong Kong, Hong Kong Island
  - Diabetes Centre, Department of Medicine and Rehabilitation, Tung Wah Eastern Hospital, Hong Kong Island
  - School of Nursing, The University of Hong Kong, Hong Kong Island

REFERENCES:
- [Result] Wong CK, Fung CS, Siu SC, Lo YY, Wong KW, Fong DY, Lam CL. A short message service (SMS) intervention to prevent diabetes in Chinese professional drivers with pre-diabetes: a pilot single-blinded randomized controlled trial. Diabetes Res Clin Pract. 2013 Dec;102(3):158-66. doi: 10.1016/j.diabres.2013.10.002. PMID 24466598
- [Derived] Wong CKH, Siu SC, Wong KW, Yu EYT, Lam CLK. Five-year effectiveness of short messaging service (SMS) for pre-diabetes. BMC Res Notes. 2018 Oct 10;11(1):709. doi: 10.1186/s13104-018-3810-y. PMID 30309382
- [Derived] Wong CK, Jiao FF, Siu SC, Fung CS, Fong DY, Wong KW, Yu EY, Lo YY, Lam CL. Cost-Effectiveness of a Short Message Service Intervention to Prevent Type 2 Diabetes from Impaired Glucose Tolerance. J Diabetes Res. 2016;2016:1219581. doi: 10.1155/2016/1219581. Epub 2015 Dec 21. PMID 26798647